CLINICAL TRIAL: NCT05514457
Title: Assessment of Visual Dyslexia Remediation Protocols - Dyslexia REMEDIATION
Acronym: Dyslexie REMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL21_0736
Record Dates: First submitted 2022-08-05; First posted 2022-08-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Dyslexia
Keywords: Dyslexia; Remediation; Visual attention span; Visual search
MeSH Terms: conditions — Dyslexia | interventions — Photic Stimulation; Protein-Arginine Deiminases; Light

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remediation group 1 (Experimental): dyslexic children
  Interventions: Behavioral: visual stimulation with I pad
- remediation group 2 (Experimental): dyslexic children
  Interventions: Behavioral: visual stimulation with lamp

INTERVENTIONS:
Behavioral: visual stimulation with I pad — At the beginning of the study, for baseline condition, children will do 4 tests (visuo-spatial perception test, visual attention span, visual research, phonology tests).
  In the first group of the study, the children will do visual research exercises on I pad 10 minutes per day during one month = remediation. They will also do 4 reading aloud tests, once a month, for 3 months. The remediation exercises will be realized during the first, second or third month.
  Arms: remediation group 1
Behavioral: visual stimulation with lamp — At the beginning of the study, for baseline condition, children will do the 4 tests like group 1.
  In the second group of the study, the children will do reading aloud tests, with lamp adjusted with different parameters = remediation (passive visual stimulation of a specific frequency believed to promote visual processing of written symbols).
  Arms: remediation group 2

SUMMARY:
Dyslexia is first described as a phonological deficit. Several studies report a neurovisual deficit in dyslexics. Some dyslexics have a visual deficit without phonological impairment, others have a pure phonological deficit, and still others have both types of deficits. From this observation the idea emerged to propose specific remediation protocols for people with visual impairments and to assess their effects on reading. At the theoretical level, if visual stimulation is able to improve reading performance, it is the demonstration of the existence of visual origin of dyslexia. At the clinical level, such a result not only opens the prospect of a different and more adapted rehabilitation for these types of dyslexia, but also the prospect, if the visual deficits are pre-existing to the learning of reading, to use them for early diagnosis and management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 8 to 12
* Diagnosed dyslexics
* Normal or corrected to normal vision
* Legal guardians of children subjects providing their free, informed and written consent to participate in the study; With the child also giving orally his consent to participate.

Exclusion Criteria:

* other neurodevelopmental problem
* strabismus, amblyopia

For the glasses (group 2) : epileptic child are excluded

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
reading performance | for arm 1: at baseline at 1 month at 2 month at 3 month For arm 2: 4 times in the same day, 4 consecutive reading sessions with a break in-between of minimum 5 minutes
  change in reading time
reading performance | for arm 1: at baseline at 1 month at 2 month at 3 month For arm 2: 4 times in the same day, 4 consecutive reading sessions with a break in-between of minimum 5 minutes
  change in number of errors

SECONDARY OUTCOMES:
score of Elementary Visuo-Spatial Perception test | one time at baseline
  comparisons of score of (lengths, sizes, angles and relative positions within and between objects). Minimum score = 36 and maximum (better) score = 72
visual attention span | one time at baseline
  number of letters identified in a single ocular fixation (200 ms)
Visual search time | one time at baseline
  average visual search time of symbols versus colored objects
performance score on the phonology tests (EVALéo 6-15 = Evaluation of written language and oral language 6-15 years) | one time at baseline
  metaphonology = removal of phonemes. Minimum score = 0 and maximum (better) score = 20

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Neurosciences de Lyon, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No